CLINICAL TRIAL: NCT03587532
Title: Assessment of Graft Perfusion and Oxygenation for Improved Outcome in Esophageal Cancer Surgery
Acronym: EDOBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Ghent (Other)
Collaborators: Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EC/2018/0671
Record Dates: First submitted 2018-06-14; First posted 2018-07-16 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Anastomotic Leak; Esophageal Cancer
Keywords: esophagectomy; indocyanine green; near infrared fluorescence
MeSH Terms: conditions — Anastomotic Leak; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Indocyanine Green Angiography (Experimental): ICG based angiography after creation of the stomach graft and after thoracic pull-up of the graft. Dynamic digital images will be obtained starting immediately after intravenous bolus administration of 0.5 mg/kg of ICG.
  Interventions: Diagnostic Test: Indocyanine green angiography; Diagnostic Test: Hemodynamic evaluation; Diagnostic Test: Biological and pathological markers of ischemia

INTERVENTIONS:
Diagnostic Test: Indocyanine green angiography — ICGA will be performed twice during standard esophagectomy: 30 minutes after the stomach graft creation and immediately before the esophagogastric anastomosis. stock dose of 25 mg ICG (Pulsion Medical Systems, Germany) will be diluted to 5 mg/mL with sterile water. An IV bolus of 0.5 mg/kg of ICG will be injected via a central venous catheter. Video data will be obtained with a charge-coupled device (CCD) camera fitted with a light-emitting diode emitting at a wavelength of 760mm (Visera® elite II, Olympus medical system corp, Tokyo, Japan). Images will be recorded starting immediately prior to injection until 3 minutes afterwards.
  Other Names: near infrared fluorescent imaging
Diagnostic Test: Hemodynamic evaluation — Advanced continuous hemodynamic monitoring during surgery will be performed using a PiCCO® (Pulse index Continuous Cardiac Output, Pulsion Medical Systems, Germany) catheter.
Diagnostic Test: Biological and pathological markers of ischemia — * Systemic and local capillary lactate on blood samples
  * Mitochondrial Respiratory activity analyses on biopsies at 3 region of interest (ROI)
  * Pathological analyses of the biopsies at 3 ROI

SUMMARY:
After the esophagectomy, the stomach is most commonly used to restore continuity of the upper gastro-intestinal tract. The esophagogastric anastomosis is prone to serious complications such as anastomotic leakage (AL) The reported incidence of AL after esophagectomy ranges from 5%-20%. The AL associated mortality ranges from 18-40% compared with an overall in-hospital mortality of 4-6%. The main cause of AL is tissue hypoxia, which results from impaired perfusion of the pedicle stomach graft. Clinical judgment is unreliable in determining anastomotic perfusion. Therefore, an objective, validated, and reproducible method to evaluate tissue perfusion at the anastomotic site is urgently needed. Indocyanine green angiography (ICGA) is a near infrared fluorescent (NIRF) perfusion imaging using indocyanine green (ICG). ICGA is a safe, easy and reproducible method for graft perfusion analysis, but it is not yet calibrated. The purpose of this study is to evaluate the feasibility of quantification of ICGA to assess graft perfusion and its influence on AL in patients after minimally invasive Ivor Lewis esophagectomy (MIE) for cancer.

DETAILED DESCRIPTION:
Background: The incidence of adenocarcinoma of the esophagus is rapidly increasing, resulting in 480 000 newly diagnosed patients annually in the world1. Surgery remains the cornerstone of therapy for curable esophageal cancer (EC) patients. After the esophagectomy, the stomach is most commonly used to restore continuity of the upper gastro-intestinal tract. The esophagogastric anastomosis is prone to serious complications such as anastomotic leakage (AL), fistula, bleeding, and stricture. The reported incidence of AL after esophagectomy ranges from 5%-20% 2-6. The AL associated mortality ranges from 18-40% compared with an overall in-hospital mortality of 4-6% 2, 7, 8. The main cause of AL is tissue hypoxia, which results from impaired perfusion of the pedicle stomach graft. Clinical judgment is unreliable in determining anastomotic perfusion. Therefore, an objective, validated, and reproducible method to evaluate tissue perfusion at the anastomotic site is urgently needed. Near infrared fluorescent (NIRF) perfusion imaging using indocyanine green (ICG) is an emerging modality based on excitation and resulting fluorescence in the near-infrared range (λ = 700-900 nm).

Aims:

* To perform intraoperative ICG based NIRF angiography of the stomach graft during minimally invasive esophagectomy in EC patients, and to calculate tissue blood flow and volume using curve analysis and advanced compartmental modeling;
* To validate imaging based perfusion parameters by comparison with hemodynamic parameters, blood and tissue expression of hypoxia induced markers, and tissue mitochondrial respiration rate
* To evaluate the ability of NIRF based perfusion measurement to predict anastomotic leakage.

Methods: Patients (N=70) with resectable EC will be recruited to undergo minimally invasive Ivor Lewis esophagectomy according to the current standard of care. ICG based angiography will be performed after creation of the stomach graft and after thoracic pull-up of the graft. Dynamic digital images will be obtained starting immediately after intravenous bolus administration of 0.5 mg/kg of ICG. The resulting images will be subjected to curve analysis (time to peak, washout time) and to compartmental analysis based on the AATH kinetic model (adiabatic approximation to tissue homogeneity, which allows to calculate blood flow, blood volume, vascular heterogeneity, and vascular leakage). The calculated perfusion parameters will be compared to intraoperative hemodynamic data (PiCCO catheter) to evaluate how patient hemodynamics affect graft perfusion. To verify whether graft perfusion truly represents tissue oxygenation, perfusion parameters will be compared with systemic lactate as well as serosal lactate from the stomach graft. In addition, perfusion parameters will be compared to tissue expression of hypoxia related markers and mitochondrial chain respiratory rate as measured in tissue samples from the stomach graft.

Finally, the ability of functional, histological, and cellular perfusion and oxygenation parameters to predict anastomotic leakage and postoperative morbidity in general will be evaluated using the appropriate univariate and multivariate statistical analyses.

Relevance: The results of this project may lead to a novel, reproducible, and minimally invasive method to objectively assess perioperative anastomotic perfusion during EC surgery. Such a tool may help to reduce the incidence of AL and its associated severe morbidity and mortality

ELIGIBILITY:
Inclusion Criteria:

Pre- and intraoperatively

* Subjects ≥ 18 years and ≤ 75 years who are willing to participate and provide written informed consent prior to any study-related procedures.
* Subjects scheduled for elective minimally invasive Ivor Lewis esophagectomy
* Intrathoracic circular stapled esophago-gastric anastomosis

Exclusion Criteria:

Preoperatively

* Known hypersensitivity to ICG
* Female patients who are pregnant or nursing
* Participation in other studies involving investigational drugs or devices.
* Use of Avastin™ (bevacizumab) or other anti vascular endothelial growth factor (VEGF) agents within 30 days prior to surgery

Intra-operatively

* Intra-operative findings that may preclude conduct of the study procedures
* Anastomosis performed differently than the standard of care
* Excessive bleeding (>500 ml) prior to anastomosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
An ICGA based cutoff point to predict anastomotic leakage and graft necrosis after esophageal reconstructive surgery. | within 3 months after intervention
  quantitative analysis of the ICGA images. T inflow will be calculated based on time fluorescence curves, and correlated with anastomotic leakage and graft necrosis. This cutoff value will be an ICGA fluorescent intensity time measurement expressed in seconds.

SECONDARY OUTCOMES:
The evaluation of ICGA as a quantitative perfusion imaging modality during gastric tube reconstruction. | within 3 months after intervention
  First, intensity over time curves will be analysed in the regions of interest to generate quantitative values for maximal fluorescence intensity (I max), inflow time (T inflow), and outflow time (T outflow). For every patient a time intensity curve will be created and From that curve 3 quantitaive time measures will be extracted: for maximal fluorescence intensity (I max), inflow time (T inflow), and outflow time (T outflow). These 3 times will be expressed in seconds
Systemic lactate as a Biological Markers of hypoxia and ischemia | within 24 hours after intervention
  Peroperative blood samples will be collected and analyzed
Capillary lactate as a Biological Markers of hypoxia and ischemia | within 24 hours after intervention
  Peroperative blood samples will be collected and analyzed
Basal oxygen consumption (V0) as a Biological Markers of hypoxia and ischemia | within 24 hours after intervention
  Peroperative biopsies will be collected and analyzed
Max respiratory oxygen consumption (Vmax) as a Biological Markers of hypoxia and ischemia | within 24 hours after intervention
  Peroperative biopsies will be collected and analyzed
Severity of inflammation score as a pathological Markers of hypoxia and ischemia | within 10 days after intervention
  Peroperative biopsies will be collected and analyzed. Four sections of the embedded material are examined using a Haematoxylin-eosin staining. A semiquantitive scoring based on presence of fibroblasts, polynuclear neutrophils, lymphocytes and macrophages will be used to evaluate the severity of the inflammation. Scoring system.
  Score 0 = normal mucosa Score 1: partial epithelial edema and necrosis Score 2: diffuse swelling and necrosis of the epithelium Score 3: necrosis with submucosal neutrophil infiltration Score 4: widespread necrosis and massive neutrophil infiltration and bleeding
HIF 1 alpha as a pathological Markers of hypoxia and ischemia | within 10 days after intervention
  Peroperative biopsies will be collected and analyzed
Minor and major adverse events up to 30 days postoperative associated with esophagectomy | within 1 year after intervention
  All adverse events will be classified by the Clavien Dindo score and based on the ECCG international consensus for complications associated with esophagectomy guidelines.The list is a predefined by the ECCG and can be found in reference 32.
Product related adverse endpoints | within 24 hours after intervention
  * Anaphylactic adverse events (AE): discomfort, flushing, tachycardia, hypotension, dyspnoea, bronchial spasm, blushing, cardiac arrest, laryngeal spasm, and facial oedema.
  * Urticarial AE: pruritus, urticaria
  * Nausea.
  * hypereosinophilia
Intensive Care Unit (ICU) stay | within 1 year after intervention
  duration of intensive care stay expressed in days
in hospital stay | within 1 year after intervention
  duration of the in hospital stay expressed in days
cardiac output | within 24 hours after the intervention
  Advanced continuous hemodynamic monitoring during surgery will be performed using a PiCCO® (Pulse index Continuous Cardiac Output, Pulsion Medical Systems, Germany). This will provide specific perfusion measurements as cardiac output expressed in liters per minute from the Pulse contour analysis and Thermo dilution analysis.
Stroke Volume | within 24 hours after the intervention
  Advanced continuous hemodynamic monitoring during surgery will be performed using a PiCCO® (Pulse index Continuous Cardiac Output, Pulsion Medical Systems, Germany). This will provide specific perfusion measurements as Stroke Volume (SV) expressed in milliliter and stroke volume variation (SVV) to predict Volume responsivity by Pulse contour analysis and Thermo dilution analysis.
pulse pressure | within 24 hours after the intervention
  Advanced continuous hemodynamic monitoring during surgery will be performed using a PiCCO® (Pulse index Continuous Cardiac Output, Pulsion Medical Systems, Germany). This will provide specific perfusion measurements as pulse pressure (PP) expressed in millimeters of mercury (mmHg) and pulse pressure variation (PPV) to predict volume responsivity by Pulse contour analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Yves.Vannieuwenhove@uzgent.be, MD, PhD, Study Director — University Hospital, Ghent
Locations (1):
- University Hospital, Ghent, Belgium

REFERENCES:
- [Background] Kassis ES, Kosinski AS, Ross P Jr, Koppes KE, Donahue JM, Daniel VC. Predictors of anastomotic leak after esophagectomy: an analysis of the society of thoracic surgeons general thoracic database. Ann Thorac Surg. 2013 Dec;96(6):1919-26. doi: 10.1016/j.athoracsur.2013.07.119. Epub 2013 Sep 24. PMID 24075499
- [Background] Biere SS, Maas KW, Cuesta MA, van der Peet DL. Cervical or thoracic anastomosis after esophagectomy for cancer: a systematic review and meta-analysis. Dig Surg. 2011;28(1):29-35. doi: 10.1159/000322014. Epub 2011 Feb 4. PMID 21293129
- [Background] Sauvanet A, Mariette C, Thomas P, Lozac'h P, Segol P, Tiret E, Delpero JR, Collet D, Leborgne J, Pradere B, Bourgeon A, Triboulet JP. Mortality and morbidity after resection for adenocarcinoma of the gastroesophageal junction: predictive factors. J Am Coll Surg. 2005 Aug;201(2):253-62. doi: 10.1016/j.jamcollsurg.2005.02.002. PMID 16038824
- [Background] Sunpaweravong S, Ruangsin S, Laohawiriyakamol S, Mahattanobon S, Geater A. Prediction of major postoperative complications and survival for locally advanced esophageal carcinoma patients. Asian J Surg. 2012 Jul;35(3):104-9. doi: 10.1016/j.asjsur.2012.04.029. Epub 2012 Jun 6. PMID 22884266
- [Background] Haga Y, Wada Y, Takeuchi H, Ikejiri K, Ikenaga M. Prediction of anastomotic leak and its prognosis in digestive surgery. World J Surg. 2011 Apr;35(4):716-22. doi: 10.1007/s00268-010-0922-5. PMID 21184072
- [Background] Rutegard M, Lagergren P, Rouvelas I, Lagergren J. Intrathoracic anastomotic leakage and mortality after esophageal cancer resection: a population-based study. Ann Surg Oncol. 2012 Jan;19(1):99-103. doi: 10.1245/s10434-011-1926-6. Epub 2011 Jul 19. PMID 21769467
- [Background] Van Daele E, Van de Putte D, Ceelen W, Van Nieuwenhove Y, Pattyn P. Risk factors and consequences of anastomotic leakage after Ivor Lewis oesophagectomydagger. Interact Cardiovasc Thorac Surg. 2016 Jan;22(1):32-7. doi: 10.1093/icvts/ivv276. Epub 2015 Oct 3. PMID 26433973
- [Background] Wright CD, Kucharczuk JC, O'Brien SM, Grab JD, Allen MS; Society of Thoracic Surgeons General Thoracic Surgery Database. Predictors of major morbidity and mortality after esophagectomy for esophageal cancer: a Society of Thoracic Surgeons General Thoracic Surgery Database risk adjustment model. J Thorac Cardiovasc Surg. 2009 Mar;137(3):587-95; discussion 596. doi: 10.1016/j.jtcvs.2008.11.042. PMID 19258071
- [Background] Junemann-Ramirez M, Awan MY, Khan ZM, Rahamim JS. Anastomotic leakage post-esophagogastrectomy for esophageal carcinoma: retrospective analysis of predictive factors, management and influence on longterm survival in a high volume centre. Eur J Cardiothorac Surg. 2005 Jan;27(1):3-7. doi: 10.1016/j.ejcts.2004.09.018. PMID 15621463
- [Background] Markar SR, Arya S, Karthikesalingam A, Hanna GB. Technical factors that affect anastomotic integrity following esophagectomy: systematic review and meta-analysis. Ann Surg Oncol. 2013 Dec;20(13):4274-81. doi: 10.1245/s10434-013-3189-x. Epub 2013 Aug 14. PMID 23943033
- [Background] Alander JT, Kaartinen I, Laakso A, Patila T, Spillmann T, Tuchin VV, Venermo M, Valisuo P. A review of indocyanine green fluorescent imaging in surgery. Int J Biomed Imaging. 2012;2012:940585. doi: 10.1155/2012/940585. Epub 2012 Apr 22. PMID 22577366
- [Background] Milstein DMJ, Ince C, Gisbertz SS, Boateng KB, Geerts BF, Hollmann MW, van Berge Henegouwen MI, Veelo DP. Laser speckle contrast imaging identifies ischemic areas on gastric tube reconstructions following esophagectomy. Medicine (Baltimore). 2016 Jun;95(25):e3875. doi: 10.1097/MD.0000000000003875. PMID 27336874
- [Background] Linder G, Hedberg J, Bjorck M, Sundbom M. Perfusion of the gastric conduit during esophagectomy. Dis Esophagus. 2017 Jan 1;30(1):143-149. doi: 10.1111/dote.12537. PMID 27766735
- [Background] Pham TH, Perry KA, Enestvedt CK, Gareau D, Dolan JP, Sheppard BC, Jacques SL, Hunter JG. Decreased conduit perfusion measured by spectroscopy is associated with anastomotic complications. Ann Thorac Surg. 2011 Feb;91(2):380-5. doi: 10.1016/j.athoracsur.2010.10.006. PMID 21256274
- [Background] Tsekov C, Belyaev O, Tcholakov O, Tcherveniakov A. Intraoperative Doppler assessment of gastric tube perfusion in esophagogastroplasty. J Surg Res. 2006 May;132(1):98-103. doi: 10.1016/j.jss.2005.07.037. Epub 2005 Sep 12. PMID 16154594
- [Background] Koyanagi K, Ozawa S, Oguma J, Kazuno A, Yamazaki Y, Ninomiya Y, Ochiai H, Tachimori Y. Blood flow speed of the gastric conduit assessed by indocyanine green fluorescence: New predictive evaluation of anastomotic leakage after esophagectomy. Medicine (Baltimore). 2016 Jul;95(30):e4386. doi: 10.1097/MD.0000000000004386. PMID 27472732
- [Background] Zehetner J, DeMeester SR, Alicuben ET, Oh DS, Lipham JC, Hagen JA, DeMeester TR. Intraoperative Assessment of Perfusion of the Gastric Graft and Correlation With Anastomotic Leaks After Esophagectomy. Ann Surg. 2015 Jul;262(1):74-8. doi: 10.1097/SLA.0000000000000811. PMID 25029436
- [Background] Yukaya T, Saeki H, Kasagi Y, Nakashima Y, Ando K, Imamura Y, Ohgaki K, Oki E, Morita M, Maehara Y. Indocyanine Green Fluorescence Angiography for Quantitative Evaluation of Gastric Tube Perfusion in Patients Undergoing Esophagectomy. J Am Coll Surg. 2015 Aug;221(2):e37-42. doi: 10.1016/j.jamcollsurg.2015.04.022. Epub 2015 Apr 30. No abstract available. PMID 26206660
- [Background] Campbell C, Reames MK, Robinson M, Symanowski J, Salo JC. Conduit Vascular Evaluation is Associated with Reduction in Anastomotic Leak After Esophagectomy. J Gastrointest Surg. 2015 May;19(5):806-12. doi: 10.1007/s11605-015-2794-3. Epub 2015 Mar 20. PMID 25791907
- [Background] Kamiya K, Unno N, Miyazaki S, Sano M, Kikuchi H, Hiramatsu Y, Ohta M, Yamatodani T, Mineta H, Konno H. Quantitative assessment of the free jejunal graft perfusion. J Surg Res. 2015 Apr;194(2):394-399. doi: 10.1016/j.jss.2014.10.049. Epub 2014 Nov 5. PMID 25472574
- [Background] Kumagai Y, Ishiguro T, Haga N, Kuwabara K, Kawano T, Ishida H. Hemodynamics of the reconstructed gastric tube during esophagectomy: assessment of outcomes with indocyanine green fluorescence. World J Surg. 2014 Jan;38(1):138-43. doi: 10.1007/s00268-013-2237-9. PMID 24196170
- [Background] Diana M, Agnus V, Halvax P, Liu YY, Dallemagne B, Schlagowski AI, Geny B, Diemunsch P, Lindner V, Marescaux J. Intraoperative fluorescence-based enhanced reality laparoscopic real-time imaging to assess bowel perfusion at the anastomotic site in an experimental model. Br J Surg. 2015 Jan;102(2):e169-76. doi: 10.1002/bjs.9725. PMID 25627131
- [Background] Diana M, Halvax P, Dallemagne B, Nagao Y, Diemunsch P, Charles AL, Agnus V, Soler L, Demartines N, Lindner V, Geny B, Marescaux J. Real-time navigation by fluorescence-based enhanced reality for precise estimation of future anastomotic site in digestive surgery. Surg Endosc. 2014 Nov;28(11):3108-18. doi: 10.1007/s00464-014-3592-9. Epub 2014 Jun 10. PMID 24912446
- [Background] Diana M, Dallemagne B, Chung H, Nagao Y, Halvax P, Agnus V, Soler L, Lindner V, Demartines N, Diemunsch P, Geny B, Swanstrom L, Marescaux J. Probe-based confocal laser endomicroscopy and fluorescence-based enhanced reality for real-time assessment of intestinal microcirculation in a porcine model of sigmoid ischemia. Surg Endosc. 2014 Nov;28(11):3224-33. doi: 10.1007/s00464-014-3595-6. Epub 2014 Jun 17. PMID 24935199
- [Derived] Van Daele E, Van Nieuwenhove Y, Ceelen W, Vanhove C, Braeckman BP, Hoorens A, Van Limmen J, Varin O, Van de Putte D, Willaert W, Pattyn P. Assessment of graft perfusion and oxygenation for improved outcome in esophageal cancer surgery: Protocol for a single-center prospective observational study. Medicine (Baltimore). 2018 Sep;97(38):e12073. doi: 10.1097/MD.0000000000012073. PMID 30235661
- See also: Cancer Statistics, GLOBOCAN 2012: Estimated Cancer Incidence, Mortality and Prevalence Worldwide in 2012. International Agency for Research on Cancer, WHO. — http://globocan.iarc.fr